CLINICAL TRIAL: NCT02867904
Title: Efficacy of Intra-operative Subacromial Corticosteroid Injections on Surgical Outcomes After Arthroscopic Shoulder Surgery
Brief Title: Intra-Operative Corticosteroid Injection During Arthroscopic Shoulder Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: It was difficult to recruit patients to get the appropriate sample size.
Sponsor: Peter Chang (Other)
Responsible Party: Sponsor-Investigator, Peter Chang, Medical Student Researcher, University of South Dakota
Organization: University of South Dakota (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016.128
Record Dates: First submitted 2016-07-20; First posted 2016-08-16 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Arthroscopic Shoulder Surgery; Intra-articular Debridement; Subacromial Decompression; Acromioplasty; Acromioclavicular Joint Resection
MeSH Terms: interventions — Methylprednisolone; Injections; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Group A (Placebo Comparator): After arthroscopic surgery the control group (Group A) will undergo a subacromial marcaine injection (standard of care).
  Interventions: Drug: Marcaine (4ml 0.5%, injection)
- Group B (Experimental): After arthroscopic surgery the experimental group (Group B) will undergo a subacromial corticosteroid injection+marcaine.
  Interventions: Drug: Methylprednisolone (40 mg depomedrol, 1ml, injection); Drug: Marcaine (4ml 0.5%, injection)

INTERVENTIONS:
Drug: Methylprednisolone (40 mg depomedrol, 1ml, injection) — Experimental Drug
  Arms: Group B
Drug: Marcaine (4ml 0.5%, injection) — Control

SUMMARY:
The purpose of this study is to assess the efficacy of intra-operative subacromial corticosteroid injections in patients undergoing arthroscopic shoulder surgery on quality of life scores and activity level when compared to a control group.

DETAILED DESCRIPTION:
This study is designed to assess whether a subacromial injection of corticosteroids at the time of arthroscopic shoulder surgery influences quality of life scores and activity level when compared to a control group. The hypothesis is that intra-operative subacromial corticosteroid injection after arthroscopic subacromial decompression surgery will provide a more rapid improvement in quality of life scores and activity levels in the post-operative period compared with controls. The study will be a placebo-controlled, double-blind prospective study. All patients necessitating arthroscopic shoulder surgery presenting to Dr. Keith Baumgarten's clinics are eligible for participation. If the patient meets the inclusion criteria, then informed consent will be obtained for participation in this study. Each patient will undergo a standard shoulder exam to assess active range of motion and complete demographics and pre-operative patient determined outcomes surveys (1. Disabilities of the Arm, Shoulder, and Hand (DASH) 2. Simple Assessment Numeric Evaluation (SANE) 3. Western Ontario Rotator Cuff (WORC)) and the Marx shoulder activity level survey (MARX). Patients will then undergo arthroscopic shoulder surgery. After arthroscopic surgery the experimental group will undergo a subacromial corticosteroid injection + marcaine while the control group will undergo a subacromial marcaine injection. Outcomes will be assessed using the same quality of life surveys and an activity level survey at post-operative visits at the time intervals: 2 weeks and 3 months and by U.S. mail at 5 months and 1 year. Active range of motion will be assessed at post-operative visits: 2 weeks, 6 weeks, and 3 months. Subjects that meet criteria to undergo arthroscopic shoulder surgery will be provided informed consent to receiving either a subacromial corticosteroid injection or placebo injection at the end of surgery. Patients will be expected to complete all pre- and post-operative quality of life surveys and activity level surveys. It will take less than 20 minutes to complete all listed surveys at each pre- and post-operative visit. Active range of motion will be assessed at each post-operative visit and subjects will be expected to take part in this physical examination as well. The duration of subject participation is 1 year from the date of initial surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years-old or older
* Male patients
* Female patients
* Patients able to speak and understand written English
* Patients presenting to the orthopedic institute clinic with shoulder pain and necessitating the procedure of arthroscopic shoulder surgery
* Specific arthroscopic procedures include: intra-articular debridement, decompression, acromioplasty, and acromioclavicular joint resection

Exclusion Criteria:

* Patients undergoing arthroscopic shoulder surgery that includes other interventions (i.e. rotator cuff repair; labral repair, etc)
* Patients with adhesive capsulitis
* Patients with significant cervical spine symptoms and/or pathology
* Patients having a history of receiving chronic pain treatment
* Patients who are currently pregnant or who become pregnant before surgery
* Patients who cannot speak or understand written english
* Patients who are under the age of 18 years of age
* As per exclusionary criteria if a subject is pregnant they will not be eligible for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand Survey (DASH) | 1 year

SECONDARY OUTCOMES:
Active Range of Motion of Shoulder | Pre-operatively and Post-operatively at 2 weeks, 6 weeks, and 3 months
  Change from baseline active range of motion will be assessed. Range of motion of the shoulder joint will be examined by having the patient actively flex, extend, abduct, adduct, internally rotate, and externally rotate the shoulder
Simple Assessment Numeric Evaluation (SANE) | 1 year
Western Ontario Rotator Cuff Survey (WORC) | 1 year
Marx Shoulder Activity Level Survey (MARX) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopedic Institute, Sioux Falls, South Dakota, United States

REFERENCES:
- [Background] Bhattacharjee DP, Biswas C, Haldar P, Ghosh S, Piplai G, Rudra JS. Efficacy of intraarticular dexamethasone for postoperative analgesia after arthroscopic knee surgery. J Anaesthesiol Clin Pharmacol. 2014 Jul;30(3):387-90. doi: 10.4103/0970-9185.137273. PMID 25190949
- [Background] Kim YJ, Lee GY, Kim DY, Kim CH, Baik HJ, Heo S. Dexamathasone added to levobupivacaine improves postoperative analgesia in ultrasound guided interscalene brachial plexus blockade for arthroscopic shoulder surgery. Korean J Anesthesiol. 2012 Feb;62(2):130-4. doi: 10.4097/kjae.2012.62.2.130. Epub 2012 Feb 20. PMID 22379567
- [Background] Stan T, Goodman EJ, Bravo-Fernandez C, Holbrook CR. Adding methylprednisolone to local anesthetic increases the duration of axillary block. Reg Anesth Pain Med. 2004 Jul-Aug;29(4):380-1. doi: 10.1016/j.rapm.2004.03.006. No abstract available. PMID 15305267
- [Background] Attardi B, Takimoto K, Gealy R, Severns C, Levitan ES. Glucocorticoid induced up-regulation of a pituitary K+ channel mRNA in vitro and in vivo. Recept Channels. 1993;1(4):287-93. PMID 8081726
- [Background] Singelyn FJ, Lhotel L, Fabre B. Pain relief after arthroscopic shoulder surgery: a comparison of intraarticular analgesia, suprascapular nerve block, and interscalene brachial plexus block. Anesth Analg. 2004 Aug;99(2):589-92, table of contents. doi: 10.1213/01.ANE.0000125112.83117.49. PMID 15271745
- [Background] Cancienne JM, Gwathmey FW, Werner BC. Intraoperative Corticosteroid Injection at the Time of Knee Arthroscopy Is Associated With Increased Postoperative Infection Rates in a Large Medicare Population. Arthroscopy. 2016 Jan;32(1):90-5. doi: 10.1016/j.arthro.2015.09.003. Epub 2015 Nov 6. PMID 26553960
- [Background] Arroll B, Goodyear-Smith F. Corticosteroid injections for osteoarthritis of the knee: meta-analysis. BMJ. 2004 Apr 10;328(7444):869. doi: 10.1136/bmj.38039.573970.7C. Epub 2004 Mar 23. PMID 15039276
- [Background] Koyonos L, Yanke AB, McNickle AG, Kirk SS, Kang RW, Lewis PB, Cole BJ. A randomized, prospective, double-blind study to investigate the effectiveness of adding DepoMedrol to a local anesthetic injection in postmeniscectomy patients with osteoarthritis of the knee. Am J Sports Med. 2009 Jun;37(6):1077-82. doi: 10.1177/0363546508331204. Epub 2009 Mar 11. PMID 19279226
- [Background] Highgenboten CL, Jackson AW, Meske NB. Arthroscopy of the knee. Ten-day pain profiles and corticosteroids. Am J Sports Med. 1993 Jul-Aug;21(4):503-6. doi: 10.1177/036354659302100404. PMID 8368408
- [Background] Armstrong RW, Bolding F. Septic arthritis after arthroscopy: the contributing roles of intraarticular steroids and environmental factors. Am J Infect Control. 1994 Feb;22(1):16-8. doi: 10.1016/0196-6553(94)90086-8. PMID 8172371
- [Background] Fontana C, Di Donato A, Di Giacomo G, Costantini A, De Vita A, Lancia F, Caricati A. Postoperative analgesia for arthroscopic shoulder surgery: a prospective randomized controlled study of intraarticular, subacromial injection, interscalenic brachial plexus block and intraarticular plus subacromial injection efficacy. Eur J Anaesthesiol. 2009 Aug;26(8):689-93. doi: 10.1097/eja.0b013e32832d673e. PMID 19593887
- [Background] HOLLANDER JL, BROWN EM Jr, JESSAR RA, BROWN CY. Hydrocortisone and cortisone injected into arthritic joints; comparative effects of and use of hydrocortisone as a local antiarthritic agent. J Am Med Assoc. 1951 Dec 22;147(17):1629-35. doi: 10.1001/jama.1951.03670340019005. No abstract available. PMID 14880415
- [Background] Sun Y, Chen J, Li H, Jiang J, Chen S. Steroid Injection and Nonsteroidal Anti-inflammatory Agents for Shoulder Pain: A PRISMA Systematic Review and Meta-Analysis of Randomized Controlled Trials. Medicine (Baltimore). 2015 Dec;94(50):e2216. doi: 10.1097/MD.0000000000002216. PMID 26683932
- [Background] Tandoc MN, Fan L, Kolesnikov S, Kruglov A, Nader ND. Adjuvant dexamethasone with bupivacaine prolongs the duration of interscalene block: a prospective randomized trial. J Anesth. 2011 Oct;25(5):704-9. doi: 10.1007/s00540-011-1180-x. Epub 2011 Jun 17. PMID 21681533
- [Background] Desmet M, Braems H, Reynvoet M, Plasschaert S, Van Cauwelaert J, Pottel H, Carlier S, Missant C, Van de Velde M. I.V. and perineural dexamethasone are equivalent in increasing the analgesic duration of a single-shot interscalene block with ropivacaine for shoulder surgery: a prospective, randomized, placebo-controlled study. Br J Anaesth. 2013 Sep;111(3):445-52. doi: 10.1093/bja/aet109. Epub 2013 Apr 15. PMID 23587875
- [Background] Zheng XQ, Li K, Wei YD, Tie HT, Yi XY, Huang W. Nonsteroidal anti-inflammatory drugs versus corticosteroid for treatment of shoulder pain: a systematic review and meta-analysis. Arch Phys Med Rehabil. 2014 Oct;95(10):1824-31. doi: 10.1016/j.apmr.2014.04.024. Epub 2014 May 16. PMID 24841629
- [Background] Westermann RW, Pugely AJ, Ries Z, Amendola A, Martin CT, Gao Y, Wolf BR. Causes and Predictors of 30-Day Readmission After Shoulder and Knee Arthroscopy: An Analysis of 15,167 Cases. Arthroscopy. 2015 Jun;31(6):1035-1040.e1. doi: 10.1016/j.arthro.2015.03.029. PMID 26048765
- [Background] Bjornholdt KT, Monsted PN, Soballe K, Nikolajsen L. Dexamethasone for pain after outpatient shoulder surgery: a randomised, double-blind, placebo-controlled trial. Acta Anaesthesiol Scand. 2014 Jul;58(6):751-8. doi: 10.1111/aas.12333. Epub 2014 May 13. PMID 24825530
- [Background] Hagiwara Y, Sugaya H, Takahashi N, Kawai N, Ando A, Hamada J, Itoi E. Effects of intra-articular steroid injection before pan-capsular release in patients with refractory frozen shoulder. Knee Surg Sports Traumatol Arthrosc. 2015 May;23(5):1536-1541. doi: 10.1007/s00167-014-2936-2. Epub 2014 Mar 19. PMID 24643358